CLINICAL TRIAL: NCT06759441
Title: Exploring the Effectiveness of a Suicide Ideation Prevention Program: Reframe-IT+
Acronym: Reframe-It+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Fundación Crecer y Sanar (Unknown); University of Talca (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Full Professor, Universidad de los Andes, Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FCS 202401
Record Dates: First submitted 2024-12-26; First posted 2025-01-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Suicidal Ideation; Depression; Anxiety; Hopelessness
Keywords: Suicidal Ideation; Children
MeSH Terms: conditions — Suicidal Ideation; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study has a quasi-experimental design, without a control group with pre-post intervention evaluation. This design is suitable to start the study of an intervention and its applicability to the target population, especially when it comes to interventions that have multiple components. This type of study allows determining changes in behavior before and after the intervention in the same subjects, which allows exploring possible effects of this intervention. This study hopes to generate evidence of the effectiveness of the intervention, taking into account the limitations of the generalization of these results as it is a quasi-experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Participants will receive an individual intervention (Reframe-It+) based on cognitive behavioral therapy, with a focus on problem-solving and help-seeking, which is carried out at the Educational Establishment with a trained psychologist. It consists of 13 weekly sessions of 25 minutes each, of which 5 sessions have a face-to-face component and 8 sessions have a face-to-face-digital component where students use a computer always in the company of a psychologist facilitating the program.
  Interventions: Behavioral: Reframe-It+

INTERVENTIONS:
Behavioral: Reframe-It+ — Reframe-IT+ is an individual intervention based on cognitive behavioral therapy, with a problem-solving and help-seeking approach, which is carried out at the Educational Establishment with a trained psychologist. It consists of 13 weekly sessions of 25 minutes each, of which 5 sessions have a face-to-face component and 8 sessions have a face-to-face-digital component where students use a computer always in the company of a psychologist facilitating the program.

SUMMARY:
Suicide is a leading cause of death among young people, with worldwide prevalence rates of suicidal ideation, suicidal ideation with a plan, and suicide attempts in youth aged 14-21 years. These behaviors have a significant negative impact on individuals, families, and the community at large. In Latin America, including Chile, suicide rates have increased in recent decades. Youth suicide prevention is a public health priority in Chile, although evidence-based interventions of high quality are lacking.

Secondary schools are a suitable and accessible setting for youth suicide prevention programs, with interventions that raise awareness about suicide and improve skills to reduce suicide attempts and suicidal ideation. Despite the effectiveness of interventions such as cognitive-behavioral therapy (CBT), these are less common in school settings, although digital technologies offer a potentially efficient way to implement suicide prevention programs in schools.

The Reframe-IT program is an Internet-based cognitive-behavioral therapy designed to reduce suicidal ideation in youth, supported by school wellness staff. Studies in Australia demonstrated the effectiveness and acceptability of Reframe-IT, although it is suggested that digital interventions may have a greater impact when combined with face-to-face sessions.

This study examined the acceptability and feasibility of a combined intervention that included Reframe-IT and four additional in-person sessions for adolescents in Chile. It is suggested that these combined interventions could be a promising strategy for youth suicide prevention in school settings, especially in Latin American countries where mental health support is limited.

DETAILED DESCRIPTION:
Suicide is a leading cause of death among young people and suicide-related behaviors (SRBs) are common. Worldwide, 12-month prevalence rates of suicidal ideation, suicidal ideation with a plan, and suicide attempts in youth aged 14-21 years are 15.4-18.4%, 7.9-10.9%, and 5.7-7.1%, respectively. Suicide and suicide-related behaviors have a significant negative impact on individuals' family, friends, and the broader community. It may also increase the risk of subsequent suicides in those exposed to death by suicide. In Latin America, suicide rates have increased over the past two decades, with Chile having one of the highest rates in the region (8.0/100,000 per year, 13.4 for men and 3.0 for women). Youth suicide prevention is a key public health priority in Chile, but limited high-quality, evidence-based interventions are available.

Secondary schools are an appropriate and accessible setting for youth suicide prevention programs and have been identified as a relevant prevention setting in national and international prevention strategies. Interventions implemented in school settings have a broad reach and facilitate prevention programs to support adolescents on a large scale. School-based prevention programs have been shown to increase suicide awareness and improve skills to reduce suicidal attempts and ideation. Indicated interventions focused on the application of clinical or psychosocial interventions (e.g., cognitive-behavioral therapy, CBT) for at-risk groups have been less common in school settings. However, evidence for these interventions is widely established in other contexts, and further school-based research on such programs is warranted.

Digital technologies are a potentially viable and efficient way to implement and scale up suicide prevention programs in schools. While digital suicide prevention programs have been shown to be safe and effective, only a small number of studies have relied on digital technologies in school settings. This is a missed opportunity, as research suggests that digital interventions for other mental health problems, such as depression and anxiety, are acceptable and minimize youth concerns regarding privacy, safety, stigma, and anonymity that may be associated with in-person programs. Digital programs may also reduce costs and increase accessibility to support when resource constraints may hinder access to services. This combination of factors has sparked significant international interest in finding technology-based solutions for suicide prevention.

The Reframe-IT program is an Internet-based cognitive behavioral therapy (CBT) program that aims to reduce suicidal ideation in youth. Reframe-IT's eight online modules have a unique focus on youth, and the program is distinguished by being designed to be facilitated and supported by school wellness staff. The staff support component is an important feature, as research suggests that digital programs delivered with support from clinicians have better treatment outcomes, lower dropout rates, and improved adherence. Reframe-IT was piloted in two phases in Australia. During the first phase, a case series study was conducted using pre- and post-tests, and results indicated that the program was associated with decreased suicidal thoughts, depression, and feelings of hopelessness. For the second phase, a pilot randomized controlled trial demonstrated that those who received the intervention had greater (although not statistically significant, due to being underpowered) reductions in suicidal ideation, depression, and hopelessness compared to the control group. Participants provided positive feedback on Reframe-IT in both studies, and it was not associated with any iatrogenic effects. Reframe-IT is currently part of a large randomized controlled trial in Australia.

Previous studies have shown that stand-alone digital interventions might have a lower impact than when combined with face-to-face sessions (26). One possible explanation suggests that face-to-face sessions may reinforce the therapeutic alliance, promoting adherence and efficacy in the digital intervention (27, 28). To our knowledge, no previous study has used combined interventions to reduce SRB delivered in school settings. The small body of evidence available suggests that school-based digital interventions targeting at-risk youth are a promising avenue for suicide prevention, primarily where mental health support is limited (29). It has been suggested that developing and testing this type of intervention is suitable in Latin American countries (30). The Reframe-IT program was adapted for Chilean youth to address this need. The current study examined the acceptability and feasibility of a combined intervention that included Reframe-IT plus four additional in-person sessions for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Students in first, second and third year of secondary school from educational establishments with high socioeconomic vulnerability.
* Students who attend educational establishments located in Santiago (Chile).
* Students who attend educational establishments with secondary education (first to fourth year of secondary school).
* Students who attend mixed educational establishments.
* Students who attend educational establishments with at least two courses in first, second and third year of secondary school.
* Students who attend educational establishments with at least 30 students per course.
* Students who attend educational establishments with vulnerability (≥55%), measured with the School Vulnerability Index - National Allocation System for Equality (IVE-SINAE). This index is the proportion of students in each school with high vulnerability. This index considers the following socioeconomic variables to group schools: mother's educational level, father's educational level, and total monthly household income, among others.
* Students who score high in suicidal ideation in the past month (score ≥ 3 on the Columbia-Suicide Severity Rating Scale (C-SSRS).

Exclusion Criteria:

* Students with severe depressive symptoms assessed by the PHQ-9 (>19 points).
* Students with high severity of psychotic symptoms assessed by the Community Assessment of Psychic Experiences-Positive Scale (CAPE, P15) with score ≥ 3 on items n°13 and/or n°14 and/or n°15.
* Students with suicide attempt(s) in the past month.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation Questionnaire (SIQ) | through study completion, an average of 1 year
  This is a 30-item self-report instrument designed to assess suicidal ideation in adolescents. It has high levels of internal consistency (α=.93) and test-retest reliability over four weeks (kappa=.72). We used a Spanish version previously validated in adolescents in Chile. In our sample, Cronbach's α at baseline was .90 and McDonald's ω was .91.
Columbia-Suicide Severity Rating Scale (C-SSRS) | through study completion, an average of 1 year
  The first 5 items explore the presence of suicidal ideation, intention, and planning and are assessed over the past month. The sixth item explores suicidal behavior either as preparation, initiation of a suicide attempt, or a suicide attempt itself in the last three months. Each item is answered Yes or No. It has been validated in an English-speaking population (range of internal reliability goes from α=0.73 to α=0.93) and a Spanish-speaking population (α=0.53). The total score range is from 0 to 6 points. According to the answers provided To the different items, the categories of severity of suicidal ideation are established: If the answer is "Yes" to item 1 and/or item 2 and "No" to all the other items, a slight risk is indicated. If the answer is "Yes" to item 2 and answer "Yes" only to item 3, it suggests that the risk is moderate. If the answer si "Yes" to item 2 and the answer is "Yes" to any of items 4, 5, and 6, it indicates that the risk is severe.
The Patient Health Questionnaire (PHQ-9) | through study completion, an average of 1 year
  Is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the 9 Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria from "0" (Never) to "3" (Almost every day). In Chile, it has been validated for the detection of Chilean people aged 20 years and older, with a sensitivity of 92% and a specificity of 89%, compared to the Hamilton Depression Scale. In addition, it presents a construct validity and a predictive validity concurrent with the International Classification of Diseases (ICD-10) criteria for depression. The interpretation is made by adding the total of the first 9 questions as follows: 0-4 points, no depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
The Generalized Anxiety Disorder 7 (GAD-7) | through study completion, an average of 1 year
  Is an instrument developed from the PRIME-MD diagnostic instrument. Although designed primarily as a screening and severity measure for generalized anxiety disorder, also has moderately good performance characteristics for other common anxiety disorders: panic disorder, social anxiety disorder, and posttraumatic stress disorder. It consists of 7 questions. Its score is calculated by assigning scores from 0 to 3, to response categories from "Never" to "Almost every day." It has been validated into Spanish, where a cut-off score of 10 showed adequate values of sensitivity (86.8%) and specificity (93.4%). The scale correlated significantly with Hamilton Anxiety Rating Scale (HAM-A) (0.852, p < 0.001), Hospital Anxiety and Depression Scale (HADS) (anxiety domain, 0.903, p < 0.001) and World Health Organization Disability Assessment Questionnaire (WHO-DAS II) (0.696, p < 0.001). The total GAD-7 score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cutoff points
Beck Hopelessness Scale (BHS) | through study completion, an average of 1 year
  Hopelessness is measured using the Beck Hopelessness Scale, a self-report scale with 20 true-false items. Nine are keyed "false" and 11 are keyed "true." Each response is assigned a score of 0 or 1 for each statement, and the total "hopelessness score" is the sum of the individual item scores. A cutoff score of 9 on the scale has been found to predict eventual suicide in clinical samples. Good internal consistency (α= .86) was observed in Chilean youth. In our sample at baseline, Cronbach's α was .82 and McDonald's ω was .82.
Community Assessment of Psychotic Experiences Scale (CAPE-P15) | through study completion, an average of 1 year
  This is a 15-item self-report instrument. Item responses range from 1 (never) to 5 (very often). The scale assesses three domains: paranoid ideation (PI, 5 items), bizarre experiences (EB, 7 items), and perceptual anomalies (AP, 3 items). Scores can range from 15 to 75. Higher scores indicate greater severity of Psychotic Experiences. All items are averaged for an overall measure of the trait being assessed. In a validation study of a Chilean population of adolescents between 13 and 18 years of age, the trifactorial nature of the scale was confirmed. Internal reliability for these factors was 0.779 for PI; 0.839 for EB; and 0.884 for AP.
Quality of life questionnaire for Child and Adolescent Version (Kidscreen-10 Index) | through study completion, an average of 1 year
  This instrument measures well-being and health-related quality of life. The Kidscreen-10 is a short version of the Kidscreen-52 and Kidscreen-27, where a Rasch analysis was applied to identify those items that represented a latent, unidimensional and global construct of HRQoL. Results of studies indicate that the Kidscreen-10 provides a generally valid measure of HRQoL in children and adolescents. It has 10 items, of which 2 items are answered on a response scale from 1 = Not at all to 5 = Extremely; and the other 8 items are answered on a response scale from 1 = Never to 5 = Always. It has a version for parents and another for children and adolescents. It has demonstrated good psychometric properties, as well as good internal consistency (Cronbach's alpha = 0.82) and good test-retest stability (r = 0.73; Intraclass Correlation Coefficient (ICC) = 0.72). The self-report version for adolescents will be used.
Brief Problem Solving Inventory (SPSI-R) | through study completion, an average of 1 year
  This is a 25-item self-report instrument that measures two adaptive problem-solving dimensions (positive problem orientation and rational problem solving) and three dysfunctional dimensions (negative problem orientation, impulsive/careless style, and avoidant style). Each item is rated on a 5-point scale ranging from not at all true for me (0) to extremely true for me (4). The Spanish version has the same factor structure and appropriate alpha coefficients for the five subscales (from .62 to .99), and an overall internal consistency of .90 in Chilean adolescents. In our sample at baseline, Cronbach's α was .83 and McDonald's ω was .83 on an overall scale.
The Cognitive-behavioural Therapy Skills Questionnaire (CBTSQ) | through study completion, an average of 1 year
  The Cognitive-behavioural Therapy Skills Questionnaire is used to test which components of CBT seem to be most active. This scale originally has 16 items. Respondents rate each item on a 5-point Likert scale, from 1 (I don't do this) to 5 (I always do this). The instrument measures two skills: cognitive restructuring (CR) and behavioural activation (BA) (i.e. changes in behavioural avoidance/control and changes in cognitive style). Both scales have good reliability (CR: α=0.88; BA: α=0.85). Two items refer to the evaluation of aspects related to a disease or treatment and since in this study we want to evaluate cognitive-behavioural skills, we have chosen to exclude these two items from the questionnaire, leaving a 14-item instrument. In a study whose publication is under review with a sample of adolescents between 15 and 18 years old, using the 14-item instrument, we found that the reliability was α=0.77 and ω=0.78 for BA, and α=0.80 and ω=0.81 for CR.
Emotional Regulation Questionnaire-CA (ERQ-CA) | through study completion, an average of 1 year
  Emotional regulation (ER) was measured using the Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA); Spanish version, validated in adolescents in Chile. It is a self-report scale of 10 items, which are rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). It assesses two styles of emotional regulation: Cognitive Reappraisal (CR, six items), which consists of redefining a potential emotion-provoking situation in such a way as to change its emotional impact, and Expressive Suppression (ES, four items), which consists of inhibiting the behavioral expression of emotion. It has a high level of reliability for each of the subscales: cognitive reappraisal subscale (α=0.83 and ω=0.84); the expressive suppression subscale (α=0.42 and ω=0.50).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete, MD, PhD, Principal Investigator — Universidad de Los Andes
Locations (1):
- Universidad de los Andes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Data about primary and secondary outcomes without identifiable variables such as name, date of birth, or others.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study and until five years after the end of the study.
Access Criteria: Any researchers who ask the principal investigator fot secondary analysis, data anonymized.
URL: https://www.ismeuandes.cl/

REFERENCES:
- [Background] World Health Organization. Suicide worldwide in 2019: global health estimates. Geneva: World Health Organization; 2021. Contract No.: CC BY-NC-SA 3.0 IGO.
- [Background] Van Meter AR, Knowles EA, Mintz EH. Systematic Review and Meta-analysis: International Prevalence of Suicidal Ideation and Attempt in Youth. J Am Acad Child Adolesc Psychiatry. 2023 Sep;62(9):973-986. doi: 10.1016/j.jaac.2022.07.867. Epub 2022 Dec 20. PMID 36563876
- [Background] Pitman A, Osborn D, King M, Erlangsen A. Effects of suicide bereavement on mental health and suicide risk. Lancet Psychiatry. 2014 Jun;1(1):86-94. doi: 10.1016/S2215-0366(14)70224-X. Epub 2014 Jun 4. PMID 26360405
- [Background] Hawton K, Hill NTM, Gould M, John A, Lascelles K, Robinson J. Clustering of suicides in children and adolescents. Lancet Child Adolesc Health. 2020 Jan;4(1):58-67. doi: 10.1016/S2352-4642(19)30335-9. Epub 2019 Oct 9. PMID 31606323
- [Background] Hill NTM, Robinson J, Pirkis J, Andriessen K, Krysinska K, Payne A, Boland A, Clarke A, Milner A, Witt K, Krohn S, Lampit A. Association of suicidal behavior with exposure to suicide and suicide attempt: A systematic review and multilevel meta-analysis. PLoS Med. 2020 Mar 31;17(3):e1003074. doi: 10.1371/journal.pmed.1003074. eCollection 2020 Mar. PMID 32231381
- [Background] Hill NTM, Too LS, Spittal MJ, Robinson J. Understanding the characteristics and mechanisms underlying suicide clusters in Australian youth: a comparison of cluster detection methods. Epidemiol Psychiatr Sci. 2020 Aug 6;29:e151. doi: 10.1017/S2045796020000645. PMID 32758330
- [Background] Teti GL, Rebok F, Rojas SM, Grendas L, Daray FM. Systematic review of risk factors for suicide and suicide attempt among psychiatric patients in Latin America and Caribbean. Rev Panam Salud Publica. 2014 Aug;36(2):124-33. PMID 25345534
- [Background] Ministerio de Salud. Chile. Informe de la década de mortalidad por suicidio. Santiago, Chile: Oficina de Vigilancia de Enfermedades No Transmisibles y Encuestas Poblacionales, Departamento de Epidemiología, Ministerio de Salud; 2022.
- [Background] Schilling SH, Carreno A, Tapia E, Mascayano F, Pitronello R, Santander F, Jorquera MJ, Burrone MS, Alvarado RV. Experts by Experience: Qualitative Evaluation of Adolescent Participation in the Development of a Technological Intervention to Prevent Youth Suicide in Chile. Front Psychiatry. 2021 Jan 25;11:522057. doi: 10.3389/fpsyt.2020.522057. eCollection 2020. PMID 33603681
- [Background] Robinson J, Cox G, Malone A, Williamson M, Baldwin G, Fletcher K, O'Brien M. A systematic review of school-based interventions aimed at preventing, treating, and responding to suicide- related behavior in young people. Crisis. 2013;34(3):164-82. doi: 10.1027/0227-5910/a000168. PMID 23195455
- [Background] World Health Organization. Live life: an implementation guide for suicide prevention in countries. Geneva: World Health Organization; 2021. Contract No.: CC BY-NC-SA 3.0 IGO.
- [Background] Calear AL, Christensen H, Freeman A, Fenton K, Busby Grant J, van Spijker B, Donker T. A systematic review of psychosocial suicide prevention interventions for youth. Eur Child Adolesc Psychiatry. 2016 May;25(5):467-82. doi: 10.1007/s00787-015-0783-4. Epub 2015 Oct 15. PMID 26472117
- [Background] Brann KL, Baker D, Smith-Millman MK, Watt SJ, DiOrio C. A meta-analysis of suicide prevention programs for school-aged youth. Children and Youth Services Review. 2021;121:105826.
- [Background] Wasserman D, Hoven CW, Wasserman C, Wall M, Eisenberg R, Hadlaczky G, Kelleher I, Sarchiapone M, Apter A, Balazs J, Bobes J, Brunner R, Corcoran P, Cosman D, Guillemin F, Haring C, Iosue M, Kaess M, Kahn JP, Keeley H, Musa GJ, Nemes B, Postuvan V, Saiz P, Reiter-Theil S, Varnik A, Varnik P, Carli V. School-based suicide prevention programmes: the SEYLE cluster-randomised, controlled trial. Lancet. 2015 Apr 18;385(9977):1536-44. doi: 10.1016/S0140-6736(14)61213-7. Epub 2015 Jan 9. PMID 25579833
- [Background] Singer JB, Erbacher TA, Rosen P. School-Based Suicide Prevention: A Framework for Evidence-Based Practice. School Mental Health. 2019;11(1):54-71.
- [Background] Breet E, Matooane M, Tomlinson M, Bantjes J. Systematic review and narrative synthesis of suicide prevention in high-schools and universities: a research agenda for evidence-based practice. BMC Public Health. 2021 Jun 10;21(1):1116. doi: 10.1186/s12889-021-11124-w. PMID 34112141
- [Background] Lai MH, Maniam T, Chan LF, Ravindran AV. Caught in the web: a review of web-based suicide prevention. J Med Internet Res. 2014 Jan 28;16(1):e30. doi: 10.2196/jmir.2973. PMID 24472876
- [Background] Stefanopoulou E, Hogarth H, Taylor M, Russell-Haines K, Lewis D, Larkin J. Are digital interventions effective in reducing suicidal ideation and self-harm? A systematic review. J Ment Health. 2020 Apr;29(2):207-216. doi: 10.1080/09638237.2020.1714009. Epub 2020 Jan 28. PMID 31989852
- [Background] Torok M, Han J, Baker S, Werner-Seidler A, Wong I, Larsen ME, Christensen H. Suicide prevention using self-guided digital interventions: a systematic review and meta-analysis of randomised controlled trials. Lancet Digit Health. 2020 Jan;2(1):e25-e36. doi: 10.1016/S2589-7500(19)30199-2. Epub 2019 Nov 29. PMID 33328037
- [Background] Cuijpers P, van Straten A, Andersson G. Internet-administered cognitive behavior therapy for health problems: a systematic review. J Behav Med. 2008 Apr;31(2):169-77. doi: 10.1007/s10865-007-9144-1. PMID 18165893
- [Background] Lehtimaki S, Martic J, Wahl B, Foster KT, Schwalbe N. Evidence on Digital Mental Health Interventions for Adolescents and Young People: Systematic Overview. JMIR Ment Health. 2021 Apr 29;8(4):e25847. doi: 10.2196/25847. PMID 33913817
- [Background] Robinson J, Hetrick S, Cox G, Bendall S, Yuen HP, Yung A, Pirkis J. Can an Internet-based intervention reduce suicidal ideation, depression and hopelessness among secondary school students: results from a pilot study. Early Interv Psychiatry. 2016 Feb;10(1):28-35. doi: 10.1111/eip.12137. Epub 2014 Mar 31. PMID 24684946
- [Background] Hetrick SE, Yuen HP, Bailey E, Cox GR, Templer K, Rice SM, Bendall S, Robinson J. Internet-based cognitive behavioural therapy for young people with suicide-related behaviour (Reframe-IT): a randomised controlled trial. Evid Based Ment Health. 2017 Aug;20(3):76-82. doi: 10.1136/eb-2017-102719. Epub 2017 Jul 12. PMID 28701336
- [Background] Robinson J, Hetrick S, Cox G, Bendall S, Yung A, Pirkis J. The safety and acceptability of delivering an online intervention to secondary students at risk of suicide: findings from a pilot study. Early Interv Psychiatry. 2015 Dec;9(6):498-506. doi: 10.1111/eip.12136. Epub 2014 Mar 31. PMID 24684927
- [Background] Byrne SJ, Bailey E, Lamblin M, McKay S, Pirkis J, Mihalopoulos C, Spittal MJ, Rice S, Hetrick S, Hamilton M, Yuen HP, Lee YY, Boland A, Robinson J. Study protocol for the Multimodal Approach to Preventing Suicide in Schools (MAPSS) project: a regionally based randomised trial of an integrated response to suicide risk among secondary school students. Trials. 2022 Mar 2;23(1):186. doi: 10.1186/s13063-022-06072-8. PMID 35236397
- [Background] Rasing SPA, Stikkelbroek YAJ, Bodden DHM. Is Digital Treatment the Holy Grail? Literature Review on Computerized and Blended Treatment for Depressive Disorders in Youth. Int J Environ Res Public Health. 2019 Dec 24;17(1):153. doi: 10.3390/ijerph17010153. PMID 31878249
- [Background] Garrido S, Millington C, Cheers D, Boydell K, Schubert E, Meade T, Nguyen QV. What Works and What Doesn't Work? A Systematic Review of Digital Mental Health Interventions for Depression and Anxiety in Young People. Front Psychiatry. 2019 Nov 13;10:759. doi: 10.3389/fpsyt.2019.00759. eCollection 2019. PMID 31798468
- [Background] Leavey K, Hawkins R. Is cognitive behavioural therapy effective in reducing suicidal ideation and behaviour when delivered face-to-face or via e-health? A systematic review and meta-analysis. Cogn Behav Ther. 2017 Sep;46(5):353-374. doi: 10.1080/16506073.2017.1332095. Epub 2017 Jun 16. PMID 28621202
- [Background] Mascayano F, Schilling S, Tapia E, Santander F, Burrone MS, Yang LH, Alvarado R. Using Information and Communication Technologies to Prevent Suicide Among Secondary School Students in Two Regions of Chile: A Randomized Controlled Trial. Front Psychiatry. 2018 Jun 5;9:236. doi: 10.3389/fpsyt.2018.00236. eCollection 2018. PMID 29922187
- [Background] Jimenez-Molina A, Franco P, Martinez V, Martinez P, Rojas G, Araya R. Internet-Based Interventions for the Prevention and Treatment of Mental Disorders in Latin America: A Scoping Review. Front Psychiatry. 2019 Sep 13;10:664. doi: 10.3389/fpsyt.2019.00664. eCollection 2019. PMID 31572242
- [Background] Nunez D, Gaete J, Meza D, Andaur J, Robinson J. Testing the Effectiveness of a Blended Intervention to Reduce Suicidal Ideation among School Adolescents in Chile: A Protocol for a Cluster Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Mar 26;19(7):3947. doi: 10.3390/ijerph19073947. PMID 35409630
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Argyropoulos SV, Ploubidis GB, Wright TS, Palm ME, Hood SD, Nash JR, Taylor AC, Forshall SW, Anderson IM, Nutt DJ, Potokar JP. Development and validation of the Generalized Anxiety Disorder Inventory (GADI). J Psychopharmacol. 2007 Mar;21(2):145-52. doi: 10.1177/0269881107069944. PMID 17329293
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Capra C, Kavanagh DJ, Hides L, Scott JG. Current CAPE-15: a measure of recent psychotic-like experiences and associated distress. Early Interv Psychiatry. 2017 Oct;11(5):411-417. doi: 10.1111/eip.12245. Epub 2015 May 12. PMID 25962504
- [Background] Reynolds WM. Suicidal ideation questionnaire: Professional manual. Odessa: Psychological Assessment Resources; 1988.
- [Background] D'Zurilla TJ, Chang EC, Nottingham EJ 4th, Faccini L. Social problem-solving deficits and hopelessness, depression, and suicidal risk in college students and psychiatric inpatients. J Clin Psychol. 1998 Dec;54(8):1091-107. doi: 10.1002/(sici)1097-4679(199812)54:83.0.co;2-j. PMID 9840781
- [Background] Beck AT, Steer RA. Manual for the Beck hopelessness scale. San Antonio, TX: Psychological Corporation. 1988.
- [Background] Jacob KL, Christopher MS, Neuhaus EC. Development and validation of the cognitive-behavioral therapy skills questionnaire. Behav Modif. 2011 Nov;35(6):595-618. doi: 10.1177/0145445511419254. Epub 2011 Sep 5. PMID 21893554
- [Background] Gullone E, Taffe J. The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): a psychometric evaluation. Psychol Assess. 2012 Jun;24(2):409-17. doi: 10.1037/a0025777. Epub 2011 Oct 24. PMID 22023559
- [Background] Ravens-Sieberer U, Erhart M, Rajmil L, Herdman M, Auquier P, Bruil J, Power M, Duer W, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. Reliability, construct and criterion validity of the KIDSCREEN-10 score: a short measure for children and adolescents' well-being and health-related quality of life. Qual Life Res. 2010 Dec;19(10):1487-500. doi: 10.1007/s11136-010-9706-5. Epub 2010 Jul 30. PMID 20668950
- [Background] Valdes JM, Diaz FJ, Christiansen PM, Lorca GA, Solorza FJ, Alvear M, Ramirez S, Nunez D, Araya R, Gaete J. Mental Health and Related Factors Among Undergraduate Students During SARS-CoV-2 Pandemic: A Cross-Sectional Study. Front Psychiatry. 2022 May 31;13:833263. doi: 10.3389/fpsyt.2022.833263. eCollection 2022. PMID 35711588
- [Background] Nunez D, Arias V, Vogel E, Gomez L. Internal structure of the Community Assessment of Psychic Experiences-Positive (CAPE-P15) scale: Evidence for a general factor. Schizophr Res. 2015 Jul;165(2-3):236-42. doi: 10.1016/j.schres.2015.04.018. Epub 2015 Apr 30. PMID 25935814
- [Background] Davis JM. Suicidal Ideation Questionnaire. Journal of Psychoeducational Assessment. 1992;10(3):298-301.
- [Background] Nuñez D, Villacura-Herrera C, Gaete J, Meza D, Andaur J, Robinson J. Psychometric assessment of the Suicidal Ideation Questionnaire Junior: A two-study validation in Spanish-speaking adolescents. Current Psychology. 2023.
- [Background] De La Torre MT, Morera OF, Wood JM. Measuring social problem solving using the Spanish version for Hispanics of the Social Problem Solving Inventory-Revised. Cultur Divers Ethnic Minor Psychol. 2010 Oct;16(4):501-6. doi: 10.1037/a0021372. PMID 21058813
- [Background] Crockett MA, Martinez V, Jimenez-Molina A. Subthreshold depression in adolescence: Gender differences in prevalence, clinical features, and associated factors. J Affect Disord. 2020 Jul 1;272:269-276. doi: 10.1016/j.jad.2020.03.111. Epub 2020 Apr 29. PMID 32553367
- [Background] Beck AT, Brown G, Berchick RJ, Stewart BL, Steer RA. Relationship between hopelessness and ultimate suicide: a replication with psychiatric outpatients. Am J Psychiatry. 1990 Feb;147(2):190-5. doi: 10.1176/ajp.147.2.190. PMID 2278535
- [Background] Alamo P. C, Baader M. T, Antúnez S. Z, Bagladi L. V, Bejer T. T. Escala de desesperanza de Beck como instrumento útil para detectar riesgo de suicidio en universitarios chilenos. Revista chilena de neuro-psiquiatría. 2019;57:167-75.
- [Background] Pastor MC, Lopez-Penades R, Cifre E, Moliner-Urdiales D. The Spanish Version of the Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): A Psychometric Evaluation in Early Adolescence. Span J Psychol. 2019 May 31;22:E30. doi: 10.1017/sjp.2019.30. PMID 31148532
- [Background] Villacura-Herrera C, Gaete J, Andaur J, Meza D, Robinson J, Núñez D. Evidence for validity, reliability and measurement invariance of the emotion regulation questionnaire for children and adolescents (ERQ-CA) in secondary students from Chile. Current Psychology. 2022.
- [Background] Baader T, Molina JL, Venezian S, Rojas C, Farías R, Fierro-Freixenet C, et al. Validación y utilidad de la encuesta PHQ-9 (Patient Health Questionnaire) en el diagnóstico de depresión en pacientes usuarios de atención primaria en Chile. Revista chilena de neuro-psiquiatría. 2012;50(1):10-22.
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Erhart M, Ottova V, Gaspar T, Jericek H, Schnohr C, Alikasifoglu M, Morgan A, Ravens-Sieberer U; HBSC Positive Health Focus Group. Measuring mental health and well-being of school-children in 15 European countries using the KIDSCREEN-10 Index. Int J Public Health. 2009 Sep;54 Suppl 2:160-6. doi: 10.1007/s00038-009-5407-7. PMID 19652910
- [Background] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308